CLINICAL TRIAL: NCT03505840
Title: TheValue of Placental Vascularization Indices and Placental Volume in Pregnancies With Antiphospholipid Syndrome for Prediction of Neonatal Outcome"
Brief Title: The Value of Placental Vascularization and Placental Volume in Pregnancy in APLS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aljazeera Hospital (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Alalfy, Assistant Researcher , National Research centre and Specialist of Obstetrics and Gynecology in Aljazeerah hospital, Aljazeera Hospital
Other Study IDs: vocal in placenta
Record Dates: First submitted 2018-04-13; First posted 2018-04-23 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Antiphospholipid Syndrome in Pregnancy
MeSH Terms: interventions — Ultrasonography; Echocardiography, Doppler

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- antiphospholipid group: pregnant ladies in the third trimester who have antiphospholipid syndrome
  Interventions: Diagnostic Test: Ultrasound with Doppler and 3D technology
- control group: pregnant ladies in the third trimester who have no medical disorders with pregnancy
  Interventions: Diagnostic Test: Ultrasound with Doppler and 3D technology

INTERVENTIONS:
Diagnostic Test: Ultrasound with Doppler and 3D technology — ultrasound will be made to pregnant females in 3rd trimester with doppler and 3D technology

SUMMARY:
Antiphospholipid antibodies are autoantibodies directed against phospholipid-binding proteins. Among these groups of antibodies, lupus anticoagulant (LA) and anticardiolipin antibodies (aCL)

DETAILED DESCRIPTION:
APLS can be primary when no evidence of autoimmune disease is found, or secondary to autoimmune processes like systemic lupus erythematous (SLE) in a 40% of the cases.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy.

  * Gestational age of 34-37 weeks.
  * Pregnant women with antiphospholipid syndrome

Exclusion Criteria:

* Twin or multiple pregnancies.
* Congenital fetal anomalies.
* Gestational age of less than 34.
* Gestational age of more than 37.
* Women with placental or umbilical artery anomalies.
* Antepartum hemorrhage (placental abruption, placenta previa and vasa previa).
* Posterior placenta.
* History of rupture of membrane.
* Patient refusal or fall outs.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant females with antiphospholipid syndrome
Study Population: Singleton pregnancy.
  * Gestational age of 34-37 weeks.
  * Pregnant women with antiphospholipid syndrome
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-04-24 (Actual); Primary Completion 2020-09-04 (Estimated); Study Completion 2020-10-10 (Estimated)

PRIMARY OUTCOMES:
The number of participants who will have impaired placental doppler indices | within 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, Principal Investigator — Algazeerah hospital -Location (Giza -Egypt ) and National Research centre egypt
Locations (1):
- Algazeerah, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No
The research data will be published